CLINICAL TRIAL: NCT06938724
Title: Omission of Local Therapies in Women Patients With HER2-positive or Triple-negative Breast Cancer: A Two Arm, Phase 2, Non-inferiority Trial for Surveillance in Maximum Responders to Neoadjuvant Systemic Therapy
Brief Title: Omission of Local Therapies in Women Patients With HER2-positive or Triple-negative Breast Cancer
Acronym: OLT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 246-24
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasm Malignant Female
Keywords: Surveillance for breast cancer relapses; Omission of local therapies; Omission of surgery; Omission of radiotherapy

STUDY DESIGN:
Intervention Model Description: This study is open to all patients with T1-2, N0-1, M0 HER2-positive or triple negative breast cancer, treated with neoadjuvant systemic treatment, irrespective of treatments delivered. The aim of the study is to evaluate outcome in maximum responders to neoadjuvant systemic therapies, when surgery or whole breast irradiation are alternatively omitted.
  Arm A will evaluate the omission of surgery in unifocal T1-2 clinically N0, M0 patients who will demonstrate maximum response after neoadjuvant systemic treatment (i.e. whole breast irradiation only).
  Arm B will evaluate the omission of radiotherapy in patients with complete pathological response proved by standard conservative surgical treatment (i.e. conservative surgery only).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Omission of Surgery (Experimental): Arm A will evaluate the omission of surgery in unifocal T1-2 clinically N0, M0 patients who will demonstrate maximum response after neoadjuvant systemic treatment (i.e. whole breast irradiation only).
  Interventions: Other: Omission of local therapies
- B Omission of Radiotherapy (Experimental): Arm B will evaluate the omission of radiotherapy in unifocal T1-2, N1, M0 patients with complete pathological response proved by standard conservative surgical treatment (i.e. conservative surgery only and surgical staging of axilla).
  Interventions: Other: Omission of local therapies

INTERVENTIONS:
Other: Omission of local therapies — Omission of surgery (arm A) or radiotherapy (arm B) in those patients who have had the maximum response by neoadjuvant treatments. Maximum responders are those patients with no evidence of residual disease after neoadjuvant treatment at imaging -including mammography, US evaluation and contrast imaging procedures (MRI and/or CEM)-, confirmed by VABB on marked site of ascertained lesion.
  This study is open to all patients with T1-2, N0-1, M0 HER2-positive or triple negative breast cancer, treated with neoadjuvant systemic treatment, irrespective of treatments delivered.

SUMMARY:
HER2-positive and Triple-negative are subtypes of breast cancer more sensitive to systemic therapies, where the complete pathological response rate may be higher than 50%. This gave rise to doubts about the usefulness of traditional local treatments for such responders. Omission of surgery after vacuum assisted breast biopsy (VABB) as well omission of radiotherapy after conservative surgery would now seem to be reasonable alternatives to standard care for highly selected patients, in whom systemic treatments have provided the maximum response.

DETAILED DESCRIPTION:
This is a prospective phase 2 non-randomized non-inferiority trial with two independent investigational arms. In each arm a 2-stage non-inferiority group-sequential design will be implemented; the overall sample per arm is of 76 patients, 43 of which will be recruited at the first stage. For each arm a futility evaluation is foreseen at the first stage, the results of which will be presented to an independent Data Safety and Monitoring Committee (iDSMC) (see "Statistical analyses" paragraph).

Arm A will evaluate the omission of surgery in unifocal T1-2 clinically N0, M0 patients who will demonstrate maximum response after neoadjuvant systemic treatment (i.e. whole breast irradiation only).

Arm B will evaluate the omission of radiotherapy in patients with complete pathological response proved by standard conservative surgical treatment (i.e. conservative surgery only). Patients candidate to arm A, who refuse the omission of surgery and then operated, are eligible for arm B if complete pathological response is confirmed after standard surgical treatment. Moreover, patients who refuse VABB and N1 patients with complete pathological response confirmed by partial mastectomy and surgical staging of axilla (SLNB and or TAD) are also eligible for arm B. Arm B patients must have confirmed complete pathological response by local-regional surgery. Therefore, omission of radiotherapy will be ultimately offered to a cohort of patients with T1-2, N0-1, M0 breast cancer conservatively operated, in whom complete pathological response to a neoadjuvant therapies is confirmed on the entire surgical specimen of the tumor bed and of the sampled nodes.

In each study arm non inferiority of 5-year EFS will be tested against historical data. No between arms statistical comparison is foreseen.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18y.
* Initial diagnosis of unifocal HER2-positive (regardless of HR status) or Triple-negative (HR positivity lower than 10% is allowed) T1-2, N0-1, M0 breast cancer.
* Treated with neoadjuvant systemic treatment according to the center recommendations.
* Maximum responders and/or complete pathological response proved by surgery.
* Scheduled for breast conservation.
* Giving specific informed consent.

Exclusion Criteria:

* One of the inclusion criteria missed.
* Residual ductal carcinoma in situ (DCIS) at VABB and/or surgery.
* Bilateral synchronous breast cancer.
* Previous malignancy within 5 years.
* BRCA1-2, PALB2 or p53 proven mutation carrier (VUS are exclusion criteria as well).
* Patients unable to perform regular follow up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2035-07-25 (Estimated); Study Completion 2035-07-25 (Estimated)

PRIMARY OUTCOMES:
Events-free survival (EFS) for each study arm. | 5 years
  Events considered are: local recurrence, distant metastases, or death, whichever will occur first.

SECONDARY OUTCOMES:
Time to rescue surgery | 5 years
  Delayed of treatment in case of local-regional disease reappearance

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Gennaro, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori Milan
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuerer HM, Smith BD, Krishnamurthy S, Yang WT, Valero V, Shen Y, Lin H, Lucci A, Boughey JC, White RL, Diego EJ, Rauch GM; Exceptional Responders Clinical Trials Group. Eliminating breast surgery for invasive breast cancer in exceptional responders to neoadjuvant systemic therapy: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2022 Dec;23(12):1517-1524. doi: 10.1016/S1470-2045(22)00613-1. Epub 2022 Oct 25. PMID 36306810
- [Background] van Hemert AKE, van Olmen JP, Boersma LJ, Maduro JH, Russell NS, Tol J, Engelhardt EG, Rutgers EJT, Vrancken Peeters MTFD, van Duijnhoven FH. De-ESCAlating RadioTherapy in breast cancer patients with pathologic complete response to neoadjuvant systemic therapy: DESCARTES study. Breast Cancer Res Treat. 2023 May;199(1):81-89. doi: 10.1007/s10549-023-06899-y. Epub 2023 Mar 9. PMID 36892723